CLINICAL TRIAL: NCT05999045
Title: Investigation of the Validity And Reliability of the Turkish Version of Evaluation of the Ability to Sing Easily (EASE-TR)
Brief Title: Turkish Version of Evaluation of the Ability to Sing Easily (EASE-TR)
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, MERVE OGULMUS UYSAL, Principal Investigator, Hacettepe University
Other Study IDs: EASE-TR
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Voice Fatigue
Keywords: Singing voice; Professional voice users
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- choir member: a person who sings in a choir
  Interventions: Other: Singing activity

INTERVENTIONS:
Other: Singing activity — The singing activity will involve a 1-hour performance, rehearsal, or lesson.

SUMMARY:
The aim of the study is to translate and culturally adapt the Turkish version of the EASE (EASE-TR) scale and investigate its validity and reliability.

DETAILED DESCRIPTION:
The study consists of two phases. In the first phase of the study, the scale will be translated and culturally adapted into Turkish. The second phase involves assessing participants and validating the translated scale. In this phase, participants will complete the EASE-TR and the severity part of the Vocal Tract Discomfort Scale (VTDS) before and after a 1-hour performance. One hundred choir member between the ages of 18 and 65 will be included in the study.

Both construct and criterion validity procedures will be used.Within the scope of construct validity, the "Known Groups Validity" method will be used based on variables such as experience duration, vocal training status, and the presence or absence of current vocal complaints. A comparison of pre- and post-performance EASE-TR scores will be conducted. Regarding criterion validity, the correlation between EASE scores and the severity part of the VTDS will be examined. For reliability, Cronbach's alpha and test-retest reliability will be calculated. The questionnaire will be administered a second time to 30 participants after 14 days in order to measure test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Having Turkish as mother tongue
* Singing in choir at least 6 months
* Performing at least for an hour

Exclusion Criteria:

* Having previously received voice therapy or undergone voice surgery
* Having a systematic/or neurological disorder that may affect voice quality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who sings in a professional or unprofessional choir
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Evaluation of the Ability to Sing Easily (EASE) Turkish Version score | 1-hour singing activity
  Turkish Version of Evaluation of the Ability to Sing Easily score: scoring ranges from 22 to 88 with higher score meaning worse outcome

SECONDARY OUTCOMES:
Vocal Tract Discomfort Scale (VTDS) | 1-hour singing activity
  The severity part of the Vocal Tract Discomfort Scale (VTDS): scoring ranges from 0 to 48 with higher score meaning worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ogulmus Uysal M, Esen Aydinli F, Incebay O, Besik Topcu O, Dasdogen U. Cross-Cultural Adaptation and Validation of the Turkish Version of the Evaluation of the Ability to Sing Easily (EASE-TR). J Voice. 2024 Nov 22:S0892-1997(24)00358-8. doi: 10.1016/j.jvoice.2024.10.016. Online ahead of print. PMID 39580357